CLINICAL TRIAL: NCT03174860
Title: Effect of Preoperative Diclofenac Potassium on Articaine Buccal Infitration Success in Mandibular Molars With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Diclofenac Potassium on Articaine Buccal Infitration Success
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amatallah Hussein Nasser Al-Rawhani, Postgraduate Student in Endodontic Department/ Faculty of Oral and Dental Medicine/ Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBC-CU-2016-11-167
Record Dates: First submitted 2017-05-09; First posted 2017-06-05 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Pulpitis - Irreversible; Anesthesia, Local
Keywords: Pulpitis, irreversible Pulpitis, Hot tooth; Cataflam, Diclofenac Potassium, Preoperative, Premedication, Analgesic; Local anesthesia, Articaine, Buccal infiltration
MeSH Terms: conditions — Pulpitis | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: The patients will be randomly divided into 2 groups:
  Experimental group:
  Diclofenac Potassium (50 mg, Cataflam) to be administered one hour before treatment.
  Control group:
  Placebo to be administered one hour before treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac Potassium 50mg tab (Experimental): Diclofenac Potassium 50mg (Cataflam) tablet to be administered one hour before treatment.
  Interventions: Drug: Diclofenac Potassium 50mg Tab
- Placebo (Placebo Comparator): Placebo to be administered one hour before treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Potassium 50mg Tab — A 50 mg tablet of the medication to be taken one hour before initiation of endodontic treatment.
  Other Names: Cataflam 50mg
  Arms: Diclofenac Potassium 50mg tab
Drug: Placebo — A placebo will be taken one hour before initiation of endodontic treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of preoperative Diclofenac Potassium (50 mg Cataflam) on the anesthetic success of buccal infiltration with 4% articaine with epinephrine 1:200,000 in mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of preoperative administration of Diclofenac Potassium (50 mg Cataflam) compared to placebo, one hour before treatment, on the anesthetic success of buccal infiltration with 4% articaine with epinephrine 1:200,000 in mandibular molars with symptomatic irreversible pulpitis. Patients with moderate-to-severe pre-operative pain are selected. Full medical and dental history will be obtained from all patients treated during this study by the operator. Clinical diagnosis of symptomatic irreversible pulpitis is to be confirmed. The primary outcome is success of buccal infiltration using articaine.The secondary outcomes are pain on injection. Patients will be recruited from the outpatient clinic of Endodontics at the Faculty of Oral and Dental Medicine, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active pain (moderate-to-severe) in mandibular molars.
* Patients with prolonged response to cold testing and electric pulp tester.
* Patient with the ability to understand and use pain scales.
* Patient with vital coronal pulp tissue on access.
* Patient who accept to enroll to the study.

Exclusion Criteria:

* Patients' allergies or any other contraindication to diclofenac potassium or articaine.
* Pregnant and lactating females.
* Patients having pain medication in the last 6 hours.
* Patient has more than one symptomatic mandibular tooth in the same quadrant.
* Patients with periradicular pathosis and/or radiolucency other than widened periodontal ligaments.
* Patients with active peptic ulcer and gastrointestinal disorders.
* Patients with history of bleeding problems or anticoagulant use within the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Success of articaine buccal infiltration. | Intraoperative
  Success of buccal infiltration using articaine. It will be measured using Heft-Parker visual analogue scale. The success will be considered if patient experienced no or mild pain (Heft-Parker VAS rating less than 54mm) while the failure will be considered if patient experience moderate-or-severe pain (Heft-parker VAS rating greater than 54mm) during access into dentin, access into pulp chamber or instrumentation of the canals.

SECONDARY OUTCOMES:
Pain on injection | Intraoperative
  The secondary outcome is pain on injection. It will be measured by Heft-Parker visual analogue scale during local anesthesia administration.

CONTACTS AND LOCATIONS:
Overall Officials: Amatallah H Al-Rawhani, Postgraduate, Principal Investigator — Faculty of Oral and Dental Medicine/ Cairo University.; Dr. Suzan AW Amin, PhD, Study Director — Faculty of Oral and Dental Medicine/ Cairo University.; Shaima'a Gawdat, PhD, Study Director — Faculty of Oral and Dental Medicine/ Cairo University.
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro MR, Groppo FC, Haiter-Neto F, Volpato MC, Almeida JF. 4% articaine buccal infiltration versus 2% lidocaine inferior alveolar nerve block for emergency root canal treatment in mandibular molars with irreversible pulpits: a randomized clinical study. Int Endod J. 2015 Feb;48(2):145-52. doi: 10.1111/iej.12293. Epub 2014 May 22. PMID 24702239
- [Background] Prasanna N, Subbarao CV, Gutmann JL. The efficacy of pre-operative oral medication of lornoxicam and diclofenac potassium on the success of inferior alveolar nerve block in patients with irreversible pulpitis: a double-blind, randomised controlled clinical trial. Int Endod J. 2011 Apr;44(4):330-6. doi: 10.1111/j.1365-2591.2010.01833.x. PMID 21692235